CLINICAL TRIAL: NCT06038630
Title: 129Xe Gas Exchange MRI to Visualize Cardiopulmonary Function
Brief Title: 129Xe MRI Cardiopulmonary
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00113114
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Disease; Chronic Thromboembolic Pulmonary Hypertension; Acute Pulmonary Embolism; Anemia; Polycythemia; Dyspnea
MeSH Terms: conditions — Lung Diseases, Interstitial; Anemia; Polycythemia; Dyspnea | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Transfusion and Phlebotomy Patients (Active Comparator): Individuals receiving treatment for their blood hemoglobin levels or are a healthy volunteer who is planning to donate blood.
  Interventions: Drug: Hyperpolarized Xe129
- Oxygen Administration Patients (Active Comparator): Individuals diagnosed with a chronic blood clot in their lungs and are planning on having surgery to remove it (CTEPH), or have an interstitial lung disease (ILD), or have dyspnea, or are a healthy volunteer.
  Interventions: Drug: Hyperpolarized Xe129; Other: Oxygen Administration
- Acute or Chronic Pulmonary Embolism Patients (Active Comparator): Individuals recently diagnosed with a blood clot in their lungs.
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Hyperpolarized xenon will be administered in multiple doses in volumes up to 25% of subject TLC followed by a breath hold of up to 15 seconds.
Other: Oxygen Administration — Oxygen administration
  Arms: Oxygen Administration Patients

SUMMARY:
The goal of this NIH-sponsored study is to characterize three biomarkers derived from 129Xe gas exchange MRI and to understand how they change in response to interventions.

DETAILED DESCRIPTION:
This study focuses on the markers that are derived from the interaction of 129Xe with pulmonary capillary red blood cells (RBCs). Specifically, the investigators focus on RBC transfer MRI, cardiogenic oscillations in 129Xe-RBC signal amplitude, and the 129Xe-RBC chemical shift.

In addition to healthy volunteers, the population to be studied will consist of patients scheduled to undergo either transfusion or phlebotomy, those with dyspnea, those with a physician diagnosis of interstitial lung disease (ILD), idiopathic pulmonary fibrosis (IPF), non-specific interstitial pneumonias (NSIP), chronic hypersensitivity pneumonitis (cHP), and sarcoid, as well as those with either chronic thromboembolic pulmonary hypertension (CTEPH) and acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers:

(Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial)

1. Outpatients of either gender, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol (Consent must be given before any study procedures are performed.)
3. Subject has no diagnosed pulmonary conditions
4. Subject has not smoked in the previous 5 years
5. Smoking history, if any, is less than or equal to 5 pack-years
6. No history of using other inhaled products more than 1/week for > 1 year

Inclusion Criteria for Transfusion and Phlebotomy Patients:

1. In-patient or outpatients of either sex, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol

And one of the following:

1. Patients who are scheduled to receive a red cell transfusion for anemia.
2. Patients who are scheduled to undergo therapeutic phlebotomy to treat erythrocytosis or polycythemia
3. Healthy volunteers undergoing voluntary whole blood donation (healthy volunteer inclusion criteria noted above)

Inclusion Criteria for Oxygen Administration Patients:

1. In-patient or outpatients of either sex, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol

And one of the following categories (ILD, Dyspnea, CTEPH, or Healthy):

1. Interstitial Lung Disease or Dyspnea

   * Physician diagnosis of Interstitial Lung Disease by a pulmonologist using established criteria or physician referral of patient with dyspnea

   OR
2. Chronic Thromboembolic Pulmonary Hypertension (CTEPH)

   * Patients with a diagnosis of CTEPH, defined as mean PA pressure >20 mmHg with a pulmonary vascular resistance >2 WU and pulmonary capillary wedge pressure ≤15 mmHg at right heart catheterization with evidence of chronic thromboembolic disease on clinical imaging after 3 months of anticoagulation
   * Scheduled for pulmonary thromboendoarterectomy (PTE) surgery and willing to re-turn 3-6 months after for optional follow-up scans

   OR
3. Healthy Volunteer (criteria noted above)

Inclusion Criteria for Acute or Chronic Pulmonary Embolism Patients:

1. In-patient or outpatients of either sex, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol

And one of the following categories (Acute or Chronic)

1. Acute Pulmonary Embolism

   * Patients presenting with acute PE 24-48hrs post-admission
   * Willing to return after 3-6 months of anti-coagulation therapy

   OR
2. Chronic Thromboembolic Pulmonary Hypertension (CTEPH)

   * Patients with a diagnosis of CTEPH, defined as mean PA pressure >20 mmHg with a pulmonary vascular resistance >2 WU and pulmonary capillary wedge pressure ≤15 mmHg at right heart catheterization with evidence of chronic thromboembolic disease on clinical imaging after 3 months of anticoagulation
   * Scheduled for pulmonary thromboendoarterectomy (PTE) surgery and willing to re-turn 3-6 months after for optional follow-up scans

Exclusion Criteria for All subjects:

Subjects presenting with any of the following will not be included in the trial:

1. MRI is contraindicated based on responses to MRI screening questionnaire
2. Subject is pregnant or lactating
3. Resting O2 saturation <90% with maximum supplemental O2 delivered by nasal canula
4. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
5. Subject has history of any known ventricular cardiac arrhythmia
6. Subject has history of cardiac arrest within the last year
7. Subject does not fit into 129Xe vest coil used for MRI
8. Subject cannot hold his/her breath for 10 seconds
9. Subject deemed unlikely to be able to comply with instructions during imaging
10. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in RBC to Membrane Ratio Pre and Post Transfusion or Apheresis | Up to 5 days pre/post transfusion or apheresis
  The investigators will validate the Hb (hemoglobin) correction model in anemia patients pre/post transfusion and blood donors pre/post apheresis.
Change in RBC (red blood cell) Chemical Shift After Oxygen Administration | Baseline, 1 day
  To test the effects of oxygen on 129Xe MRI/MRS in healthy subjects, those with ILD, those with dyspnea, and patients with chronic thromboembolic pulmonary hypertension (CTEPH).
Change in RBC Oscillation Amplitude Post Therapy | Baseline, 3-6 months post-treatment
  Patients with chronic PE are treated surgically and those with acute PE are treated with anticoagulation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mammarappallil, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A major focus of this work is sharing and dissemination of the image acquisition and analysis methods we develop as well as standard operating procedures for 129Xe MRI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In all instances we will adhere to the NIH Sharing Policies and Related Guidance on NIH-Funded Research Resources for Recipients of NIH Grants and Contracts on Obtaining (https://grants.nih.gov/policy/sharing.htm) and Disseminating Biomedical Research Re-sources (issued December 1999). However, we intend to greatly exceed these requirements, making as much of our work freely available to the broader research community either before, or immediately after publication of manuscripts, as well as through PubMedCentral. While we will provide relevant protocols upon request at any time, we further intend to pursue several proactive data sharing mechanisms.
Access Criteria: We are committed to making de-identified datasets and image analysis available to qualified investigators. When required scientifically, data including identifiers will be shared under an agreement that provides for: (1) a commitment to using data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data appropriately; and (3) a commitment to destroying or returning the data after analyses are completed.